CLINICAL TRIAL: NCT05108727
Title: Clinical and Microbiological Evaluation of Diode Laser- Assisted-Flap Surgery for the Treatment of Patients With Stage 3-Grade C Periodontitis: 6-month Randomized Split-mouth Clinical Trial
Brief Title: Diode Laser With Periodontal Flap Surgery in Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Seyma Bozkurt Doğan, Associate Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-21-008
Record Dates: First submitted 2021-10-24; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Periodontitis, Aggressive; Diode Laser Therapy; Periodontal Diseases
Keywords: diode laser; aggressive periodontitis; Modified Widman Flap; microbiology
MeSH Terms: conditions — Aggressive Periodontitis; Periodontal Diseases | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Diode Laser Therapy+ Modified Widman Flap (Active Comparator): Diode laser with a wavelength of 810±5 nm and a power of 1 watt in continuous mode was applied to the Modified Widman Flap at the test sites
  Interventions: Device: Diode Laser; Procedure: Modified Widman Flap
- Sham Diode Laser Therapy+ Modified Widman Flap (Sham Comparator): Control sites were treated with MWF alone
  Interventions: Procedure: Modified Widman Flap

INTERVENTIONS:
Device: Diode Laser — DL with a wavelength of 810±5 nm, a 400micron diameter, and a power of 1 watt in continuous mode was applied to the MWF at the test sites.
  Other Names: Modified Widman Flap (MFW)
  Arms: Active Diode Laser Therapy+ Modified Widman Flap
Procedure: Modified Widman Flap — Periodontal Surgery Technique

SUMMARY:
The authors theorize that periodontal flap surgery therapy with adjunctive DL therapy might bring favourable therapy results (clinical and bacterial parameters) in patients with stage 3-grade C periodontitis. Therefore, the goal of this split-mouth randomized clinical trial was to evaluate and compare the effectiveness of the treatment results for DL assisted modified Widman Flap (MWF) surgery (test site) with MWF surgery alone (control site) in periodontitis patients with stage 3-grade C by determining the changes in clinical parameters and bacterial load of pathogens (P.g., T.d., Camplyobacter rectus (C.r.), Prevotella intermedia (P.i.), T.f., A.a.) at preoperative and following MWF surgery at 6th week, 3rd and 6th months

DETAILED DESCRIPTION:
A randomised control split-mouth study were performed at the Department of Periodontology, Faculty of Dentistry, Bülent Ecevit University, Zonguldak, Turkey, between January 2013 and February 2016.After clinical evaluation, a total of 30 subjects, who showed signs of stage 3-grade C periodontitis, were enrolled to this study at baseline. These patients were underwent a full mouth scaling and root planning (SRP). Six weeks after non surgical periodontal therapy, periodontal assessment was performed to confirm the suitability of the sites for periodontal surgery. This split-mouth study was conducted in 18 patients with stage 3 Grade C periodontitis aged between 22 and 35 years.

Before the surgery, the selected quadrants were randomly allocted (by the toss of a coin) into test and control sites where the control site were treated with MWF+sham application of DL and test sites were treated with MWF+ active DL. Clinical parameters including CAL, PD, plaque index(PI), gingival index(GI), bleeding on probing (BOP) were recorded and microbiological sampling were obtained at preoperative and at 6 weeks, 3 months, 6 months postoperatively. Pain scale assessment (visual analog scale, VAS), pain medication consumption (PM), tissue edema (TE), and tissue color (TC) were evaluated one week following surgery. Microbiological analysis was done by real-time polymerase chain reaction (PCR) for detection of Porphyromonas gingivalis (P.g.), Treponema denticola (T.d.), Tannerella forsythia (T.f.), Camplyobacter rectus (C.r.), Prevotella intermedia (P.i.), Aggregatibacter actinomycetemcomitans (A.a.).

Control sites were treated MWF with sham application of DL, while test sites were treated MWF with the applying of active DL (810nm±5, Picasso-AMD, USA) to the inside of the MWF. The interval between the two surgeries was 3 weeks. The modified Widman flap technique was applied.DL with a wavelength of 810±5 nm and a power of 1 watt in continuous mode was applied to the MWF at the test sites. A 400 micron diameter tip was used to remove all visible epithelium on the inside of the flap from the free gingival edge to the lower apical aspect of the flap (both labial and lingual / palatal). The tip was started using a blue articulating paper. DL irradiation performed at a 45o angle to the soft tissue flap to avoid any laser (810nm±5) contact to the root surface or the alveolar bone . DL therapy was carried out to soft tissue from the coronal to the apical aspect in parallel paths for 10seconds. When irradiation exceeded 10 seconds in time, laser (810nm) emission was be interrupted for 30 seconds. The resultant char layer was be totally removed with moist gauze prior to replacing the flaps. A second laser application with the same laser (810nm±5) was performed on all the surfaces of the flap in continuous mode at 0.1 watts. All surfaces of the flap, inner and outer, exposed bone and exposed root structures involved in the surgery were irradiated, leading to a total dosage of 4 J/cm2 per surface.

The subjects were prescribed 200 mg Ibuprofen (up to 3 tablets) every 8 hours to reduce pain. The subjects were instructed not to eat solid food using the treated area and to not brush the teeth in the treated area. They were told to rinse their mouth with chlorhexidine digluconate (0.2%, CHX) twice a day for 1 min during one week after surgery The sutures were removed at first week . After 1 weeks, the subject started brushing their teeth and oral hygiene training was repeated. Oral hygiene instructions were provided at each postoperative visit.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for stage 3-grade C periodontitis patients were interdental CAL ≥ 5 mm and PD ≥ 6 mm on at least 6 teeth and at least three of these six teeth were not molars or incisors.
* They were under 35 years of age.
* These patients had at least two quadrants of maxilla with three teeth each having CAL ≥ 5 mm and PD ≥ 6 mm.

Exclusion Criteria:

* : systemic conditions such as; diabetes mellitus, cancer, cardiovascular and respiratory diseases,
* current and ex-smoking habits,
* undergone non-surgical periodontal therapy and prescription of antibiotics or non-steroidal anti-inflammatory medication within the previous 6 months or surgical periodontal treatment within the preceding year,
* pregnancy, lactation, postmenopause, or immunologic disorders,

Ages: 22 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level | 6 months
  distance between the cemento-enamel junction to the deepest point of periodontal pocket

SECONDARY OUTCOMES:
Probing depth | 6 months
  distance between the gingival margin to the deepest point of periodontal pocket

OTHER OUTCOMES:
Plaque index | 6 months
  oral hygiene scores: 0: no plague, 3: visible plaque
Gingival index | 6 months
  gingival inflammation score 0: no bleeding, 3: severe bleeding
Counts of bacteria | 6 months
  change in bacteria levels
Vascular analog scale | postoperatively first week
  Pain scale: 1: no pain 10: severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Figen Öngöz Dede, PhD, DDS, Principal Investigator — Ordu University; Şeyma Bozkurt Dogan, PhD, DDS, Study Chair — Ankara Yildirim Beyazıt University

REFERENCES:
- [Derived] Dogan SB, Akca G. Clinical Evaluation of Diode Laser-Assisted Surgical Periodontal Therapy: A Randomized Split-Mouth Clinical Trial and Bacteriological Study. Photobiomodul Photomed Laser Surg. 2022 Sep;40(9):646-655. doi: 10.1089/photob.2022.0035. Epub 2022 Sep 7. PMID 36070584